CLINICAL TRIAL: NCT00537134
Title: Safety and Efficacy of Endovascular Treatment of Unruptured Intracranial Aneurysms in the Prevention of Aneurysmal Haemorrhages: A Randomized Comparison With Indefinite Deferral of Treatment in 2002 Patients Followed for 10 Years
Brief Title: Trial on Endovascular Aneurysm Management
Acronym: TEAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The CIHR Financial support was withdrawn because of insufficient recruitment.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCT-80799; ISRCTN62758344 (Registry Identifier: primary clinical trial registry recognised by WHO and ICMJE)
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Brain Aneurysm
Keywords: Aneurysm; Brain; Unruptured; observation; treatment; Endovascular
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm | interventions — Embolization, Therapeutic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative (No Intervention): Conservative management (watchful observation)
- Endovascular (Active Comparator): Endovascular treatment
  Interventions: Device: Embolization, coiling

INTERVENTIONS:
Device: Embolization, coiling — Endovascular embolization with platinum coils
  Other Names: Standard and bioactive coils
  Arms: Endovascular

SUMMARY:
The management of patients with unruptured aneurysms is controversial. Patients with unruptured aneurysms may suffer intracranial hemorrhage, but the incidence of this event is still debated. Endovascular treatment can prevent rupture, but involves immediate risks; furthermore, successful treatment does not eliminate all risks. A randomized trial may be the best way to demonstrate the potential benefits of endovascular over conservative management of unruptured aneurysms.

DETAILED DESCRIPTION:
This study is designed as a pragmatic trial. All candidates for endovascular treatment of one or more unruptured intracranial aneurysms will be offered to participate. Unruptured aneurysms may be recently discovered or prevalent. If they accept, subjects will be randomized to one of the two arms of the trial: Conservative management (Observation) or Endovascular treatment.

Both groups will be advised to obtain medical treatment for hypertension if necessary and will receive counselling for behavioural risk factor modelling (smoking or excessive drinking) when indicated. A non-invasive (MRA or CTA) or catheter angiogram and a baseline CT-scan or MRI of the brain are required to enter the study. These studies should demonstrate the unequivocal presence of a saccular aneurysm >=3 mm treatable by endovascular methods. A catheter angiogram is required if there is doubt. Imaging studies will be reviewed centrally. Both treatments will be standardized. Patients will be followed similarly for a minimum of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* At least one documented subarachnoid aneurysm, never ruptured
* Patient aged 18 or older
* Life expectancy more than 10 years

Exclusion Criteria:

* Patients with recent (less than 3 months) intracranial haemorrhage
* Lesion characteristics unsuitable for endovascular treatment
* Patients with a single extradural aneurysm
* Aneurysms < 3 mm or giant aneurysms (≥ 25 mm)
* Patients with a poor outcome (Rankin scale ≥ 3) after the rupture, surgical or endovascular treatment of another aneurysm
* Patients with incompletely treated aneurysms that have previously ruptured
* Patients with associated arteriovenous malformations
* Patients with new severe progressive symptoms in relationship with the aneurysm (sudden onset, severe persisting headaches suggestive of impending rupture, third-nerve palsy, mass-effect)
* Patients with previous intracranial haemorrhage from unknown etiology
* Patients with multiple unruptured aneurysms in whom surgical clipping of one or many aneurysms is planned in addition to endovascular management
* Patients with absolute contraindications to anaesthesia, endovascular treatment, or administration of contrast material, including low-osmolarity agents or gadolinium
* Pregnant patients
* Patients unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2009-06-28 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Raymond, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal - Hôpital Notre-Dame; Andrew J. Molyneux, MD, Principal Investigator — NRU, Radcliffe Infirmary Oxford University UK; Allan J Fox, MD, Principal Investigator — Sunnybrook Health Sciences Centre and University of Toronto; Claiborne S. Johnston, MD, PhD, Principal Investigator — University of California, San Francisco, USA; Jean-Paul Collet, MD, PhD, Principal Investigator — University of British Columbia, Vancouver, Canada; Isabelle Rouleau, PhD, Principal Investigator — CHUM Hôpital Notre-Dame, Montreal, Canada
Locations (9):
- United States (6):
  - St Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Boston Medical Center, Boston, Massachusetts
  - SUNY Downstate Medical Center, Brooklyn, New York
  - St Luke's-Roosevelt Hospital Center, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - The Methodist Hospital, Houston, Texas
- CHUM Notre-Dame Hospital / TEAM clinical research unit (Head office), Montreal, Quebec, Canada
- TEAM France Coordination Unit - CHU Reims CRICAM, Reims, France
- TEAM European Coordination Centre NVRU- Radcliffe Infirmary, Oxford, United Kingdom

REFERENCES:
- [Background] Raymond J, Meder JF, Molyneux AJ, Fox AJ, Johnston SC, Collet JP, Rouleau I; Trial on Endovascular Aneurysm Management (TEAM) collaborative group. Trial on endovascular treatment of unruptured aneurysms (TEAM): study monitoring and rationale for trial interruption or continuation. J Neuroradiol. 2007 Mar;34(1):33-41. doi: 10.1016/j.neurad.2007.01.011. PMID 17316800
- [Background] Raymond J, Meder JF, Molyneux AJ, Fox AJ, Johnston SC, Collet JP, Rouleau I; Trial On Endovascular Aneurysm Management Team Collaborative Group. Unruptured intracranial aneurysms: the unreliability of clinical judgment, the necessity for evidence, and reasons to participate in a randomized trial. J Neuroradiol. 2006 Oct;33(4):211-9. doi: 10.1016/s0150-9861(06)77266-2. No abstract available. PMID 17041525
- [Background] Raymond J, Guilbert F, Weill A, Roy D. Unruptured intracranial aneurysms: a call for a randomized clinical trial. AJNR Am J Neuroradiol. 2006 Feb;27(2):242-3. No abstract available. PMID 16484380
- [Background] Raymond J, Guilbert F, Weill A, Georganos SA, Juravsky L, Lambert A, Lamoureux J, Chagnon M, Roy D. Long-term angiographic recurrences after selective endovascular treatment of aneurysms with detachable coils. Stroke. 2003 Jun;34(6):1398-403. doi: 10.1161/01.STR.0000073841.88563.E9. Epub 2003 May 29. PMID 12775880
- [Background] Raymond J, Chagnon M, Collet JP, Guilbert F, Weill A, Roy D. A randomized trial on the safety and efficacy of endovascular treatment of unruptured intracranial aneurysms is feasible. Interv Neuroradiol. 2004 Jun 29;10(2):103-12. doi: 10.1177/159101990401000202. Epub 2004 Oct 22. PMID 20587222
- [Background] Raymond J, Molyneux AJ, Fox AJ, Johnston SC, Collet JP, Rouleau I; TEAM Collaborative Group. The TEAM trial: safety and efficacy of endovascular treatment of unruptured intracranial aneurysms in the prevention of aneurysmal hemorrhages: a randomized comparison with indefinite deferral of treatment in 2002 patients followed for 10 years. Trials. 2008 Jul 16;9:43. doi: 10.1186/1745-6215-9-43. PMID 18631395
- [Derived] Naggara O, Raymond J, Guilbert F, Roy D, Weill A, Altman DG. Analysis by categorizing or dichotomizing continuous variables is inadvisable: an example from the natural history of unruptured aneurysms. AJNR Am J Neuroradiol. 2011 Mar;32(3):437-40. doi: 10.3174/ajnr.A2425. Epub 2011 Feb 17. PMID 21330400
- [Derived] Raymond J. Incidental intracranial aneurysms: rationale for treatment. Curr Opin Neurol. 2009 Feb;22(1):96-102. doi: 10.1097/wco.0b013e32831fee91. PMID 19165956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants are recruited when seen in clinic either for neurological symptoms or when aneurysm is an incidental finding
Pre-assignment Details: there are no pre-assignment procedures before assignment to groups
Groups:
- Endovascular: Endovascular treatment by coil embolization
  Embolization, coiling: Endovascular embolization with platinum coils
Period: Overall Study
Arm/Group | Endovascular | Conservative
Started | 42 | 38
Completed | 42 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Conservative: Conservative management (watchful observation)
  Inclusion criteria:
  1. At least one documented subarachnoid aneurysm, never ruptured
  2. Patient aged 18 or older
  3. Life expectancy more than 10 years
  Exclusion crieria:
  1. Patients with recent (less than 3 months) intracranial haemorrhage
  2. Lesion characteristics unsuitable for endovascular treatment
  3. Patients with a single extradural aneurysm
  4. Aneurysms <3mm or giant aneurysms (≥25mm)
  5. Patients with a poor outcome (Rankin scale ≥3) after the rupture, surgical or endovascular treatment of another aneurysm
  6. Patients with incompletely treated aneurysms that have previously ruptured
  7. Patients with associated arteriovenous malformations
  8. Patients with new severe progressive symptoms in relationship with the aneurysm (sudden onset, severe persisting headaches suggestive of impending rupture, third-nerve palsy, mass-effect)
  9. Patients with previous intracranial haemorrhage from unknown aetiology
  10. Patients with multiple unruptured aneurysms in whom surgical clipping of one or many aneurysms is planned in addition to endovascular management
  11. Patients with absolute contraindications to anaesthesia, endovascular treatment, or administration of contrast material, including low-osmolarity agents or gadolinium
  12. Pregnant patients
  13. Patients unable to give informed consent
- Endovascular: Endovascular treatment
  Embolization, coiling: Endovascular embolization with platinum coils
  Same population as Conservative management
- Total: Total of all reporting groups
Arm/Group | Conservative | Endovascular | Total
Number analyzed (Participants) | 38 | 42 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 63
  >=65 years | 7 | 10 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 11 | 17 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 20 | 31
  United States | 3 | 1 | 4
  United Kingdom | 9 | 9 | 18
  France | 11 | 10 | 21
  Poland | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease or Treatment-related Morbidity and Mortality.
Description: Morbidity or mortality is evaluated using the modified Rankin Scale (mRS) which goes from 0 to 6, with 0 for no symptoms at all, and 6 for Mortality. The scores were attributed using a structured interview process.
  a "Good" Primary Outcome was categorized from mRS scores of 0, 1, or 2. a "Bad" Primary Outcome was categorized from mRS scores of 3, 4, 5 or 6.
Time Frame: 1 year after treatment or observation
Measure: Count of Participants; unit: Participants
Arm/Group | Conservative | Endovascular
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

2. Secondary Outcome: Rate of Hemorrhage in Conservative Group
Description: To better define the natural history of unruptured aneurysms eligible for endovascular treatment.
Time Frame: At 5 and 10 years
Population: No patients available for outcome measure at 5 years because study was terminated
Arm/Group | Conservative | Endovascular
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Hemorrhage in Endovascular Group
Description: Number of participants experiencing a hemorrhagic event despite successful treatment.
  This outcome measure gives an estimate of risk of rupture despite treatment
Time Frame: At 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Conservative | Endovascular
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

4. Secondary Outcome: Number of Participants in Each Score of the Modified Rankin Scale in Endovascular Group
Description: The modified Rankin Scale (mRS) goes from 0 to 6, with 0 for no symptoms at all, and 6 for Mortality. The scores were attributed using a structured interview process.
  The number of participants having in each score is given.
Time Frame: At 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Conservative | Endovascular
Number analyzed (Participants) | 12 | 11
Participants
  mRS is 0 | 10 | 8
  mRS is 1 | 2 | 2
  mRS is 2 | 0 | 1

5. Secondary Outcome: Modified Rankin Score
Description: To compare overall Morbidity/Mortality of the 2 groups
Time Frame: At 10 years
Population: No patients available for outcome measure at 10 years because study was terminated
Arm/Group | Conservative | Endovascular
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Measures on 36-Item Short-Form Health Survey (SF-36)
Description: To compare the quality of life and anxiety levels of surviving patients of the 2 groups according to the SF-36 questionnaire minimum is 0 (maximum disability) maximum is 100 (No disability)
Time Frame: At 5 and 10 years
Population: No patients available for outcome measure at 5 and 10 years because study was terminated
Arm/Group | Conservative | Endovascular
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Occlusion State in the Endovascular Group
Description: To determine the rate of occlusion of aneurysms treated by coiling in an effort to estimate longer-term efficacy.
Time Frame: At 5 and 10 years
Population: No patients available for outcome measure at 5 years because study was terminated
Arm/Group | Conservative | Endovascular
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Occlusion State of the Aneurysm in the Conservative Group
Description: To determine the rate of aneurysmal growth in the conservative group in surviving patients.
Time Frame: At 5 and 10 years
Population: No patients available for outcome measure at 5 years because study was terminated
Arm/Group | Conservative | Endovascular
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With a "Bad" Cognitive Function Evaluated According to the Montreal Cognitive Assessment Scale (MoCA)
Description: To verify cognitive functions using the MoCA in all patients before and 6 months after treatment in a consecutive sample of 100 patients of both groups.
  Minimum value on the MoCA is 0 (maximum cognitive decline) Maximum value on the MoCA is 30 (no cognitive decline) A score higher than 26 was categorized as "good" cognitive condition A score of 26 or lower was categorized as "bad" cognitive conditionn
Time Frame: Baseline, 1 year, 5 and 10 years
Population: Patients with MoCa scores at Baseline and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Conservative | Endovascular
Number analyzed (Participants) | 11 | 9
Participants
  Baseline: Score is 26 or lower | 1 | 4
  Baseline: Score is higher than 26 | 10 | 5
  1 year: Score is 26 or lower | 3 | 2
  1 year: Score is higher than 26 | 8 | 7

ADVERSE EVENTS:
Time Frame: The number of patients in each period of time over which Adverse event data was collected is variable, because the study was terminated while patients were at variable points through their expected follow-up period. For example, only 52/80 participants were evaluated at 1 month before the study was terminated; at each subsequent time point, fewer participants were evaluated. - 3 years: 2 patients - 2 years: 11 patients - 1 year: 25 patients - 6 months: 41 patients - 1 month: 52 patients
Description: The definition of adverse event does not differ from the ClinicalTrials.gov definition
Arm/Group | Conservative | Endovascular
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/42
Other Adverse Events (participants affected / at risk) | 2/38 | 3/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conservative (N=38) | Endovascular (N=42)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conservative (N=38) | Endovascular (N=42)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Migraine (General disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
arm hematoma (Surgical and medical procedures) | 0 (0) | 1 (1) — hematoma resulting from arm arterial line complication

LIMITATIONS AND CAVEATS:
No conclusions can be drawn from the reported results because the study, projected to follow patients for 10 years was terminated by the funding agency after 3 years

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Statistical Analysis Plan (2007-03-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT00537134/SAP_000.pdf